CLINICAL TRIAL: NCT05249634
Title: Effect of JATENZO® Therapy on Testosterone and Hemoglobin Concentrations in Hypogonadal Men with Chronic Kidney Disease
Brief Title: Testosterone Treatment in Men with Chronic Kidney Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Louis University (Other)
Collaborators: Clarus Therapeutics, Inc. (Industry)
Responsible Party: Principal Investigator, Sandeep Singh Dhindsa, M.D., Professor of Medicine, St. Louis University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 32358
Record Dates: First submitted 2022-02-01; First posted 2022-02-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hypogonadism, Male; Kidney Disease, Chronic
Keywords: testosterone; CKD
MeSH Terms: conditions — Eunuchism; Renal Insufficiency, Chronic | interventions — Testosterone Propionate; Testosterone

STUDY DESIGN:
Intervention Model Description: All subjects will receive treatment with JATENZO
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment (Experimental): JATENZO daily for 6 months
  Interventions: Drug: Jatenzo Pill

INTERVENTIONS:
Drug: Jatenzo Pill — oral tablet daily
  Other Names: oral testosterone

SUMMARY:
This study in being conducted in men who have low testosterone and chronic kidney disease. The investigators will evaluate the effects of an oral testosterone preparation, JATENZO, on testosterone levels and hemoglobin (red blood cells).

DETAILED DESCRIPTION:
* Purpose. The purpose of this research is to find out if JATENZO will help increase testosterone levels in men with hypogonadism and chronic kidney disease, determine if there is any improvement in testosterone levels, hemoglobin (red blood cells), muscle strength, lean mass and sexual function.
* The dug will be daily for 6 months. Study Procedures. Every 2-4 weeks, the study participant will come in person for a research visit. Investigators will collect a blood sample at certain visits, do a brief physical exam, and obtain vital signs such as height, weight, blood pressure. The study also involves completing questionnaires, measuring body composition by a scan and testing muscle strength. The dose of JATENZO may be adjusted based on the testosterone levels.

ELIGIBILITY:
Inclusion Criteria:

* Men between ages of 18-85 years of age
* eGFR 15-45 ml/min/1.73m2 by MDRD (Modification of Diet in Renal Disease) equation
* Subnormal total serum T concentrations (<300 ng/dl) on two separate occasions in morning
* Symptoms of hypogonadism (as per Endocrine Society guidelines): low libido, erectile dysfunction, fatigue, irritability, depressed mood, poor concentration, increased body fat, decreased muscle bulk, reduced physical performance, sleep disturbance, loss of body hair (15)
* Normal iron stores as defined by serum ferritin ≥100 ng/mL and transferrin saturation (TSAT) ≥20%.

Exclusion Criteria:

* Use of TRT currently or in the past 6 months, including use of over-the-counter androgen containing health supplements (e.g., DHEA)
* Hematocrit >48% (as per Endocrine Society guidelines)(15)
* Treatment with erythropoiesis stimulating agents (ESA)
* Uncontrolled blood pressure (>180/100 mm Hg)
* Heart Failure, class III or IV
* Myocardial infarction, stroke, or heart surgery in the past 3 months
* Breast cancer
* History of prostate cancer
* Prostate specific antigen (PSA) >4 ng/ml, unless prostate cancer has been ruled out by a urologist (documented in physician notes)
* HIV or untreated hepatitis C
* Untreated, severe obstructive sleep apnea
* Initiated iron replacement in the last 3 months
* deep venous thrombosis or pulmonary embolism in the last 3 months
* recurrent (more than once) deep venous thrombosis or pulmonary embolism
* use of warfarin
* Planning to have children in the next one year

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Testosterone concentrations | 6 months
  Testosterone concentrations in serum measured multiple times during the study

SECONDARY OUTCOMES:
Hemoglobin | 6 months
  blood test
muscle strength | 6 months
  Hand-grip strength will be measured by a quantitative handgrip dynamometer in the dominant arm. Mean of three consecutive measurements will be used.
Lean mass | 6 months
  measured by DEXA scan
sexual function | 6 months
  Psychosexual daily questionnaire for 7 consecutive days will be used. The questionnaire covers three different domains: 1) sexual desire, enjoyment, and performance; 2) sexual activity score; and 3) mood. Sexual desire (question 1) and sexual enjoyment (question 2) will be rated on a 7-point Likert-type scale from 0 to 7, with 0 indicating none and 7 indicating very high. Sexual performance will be assessed by % full erection and satisfaction with erection (questions 5 and 6). Sexual activity (question 4) will be assessed using a checklist format. The value will be recorded as 0 (none) or 1 (any) for analysis. Higher score indicates higher activity; maximum score on this item is 12. Each mood parameter (question 3) will also be assessed on the 7-point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Dhindsa, MD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis Univeristy, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No